CLINICAL TRIAL: NCT01348828
Title: Prospective, Multicenter, Single Arm Feasibility and Safety Study of the Endologix Fenestrated Stent Graft System for the Endovascular Repair of Juxtarenal/Pararenal (JAA/PAA) Aneurysms
Brief Title: Feasibility and Safety Study of the Endologix Fenestrated Stent Graft System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-0003
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; Fenestrated; Renal Stent; Juxtarenal; Pararenal; Endologix; Renal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Other): All patients meet study criteria receives a single use Ventana Fenestrated System, which requires administration of intravascular contrast. Catheter advancement is performed under fluoroscopic guidance and Ventana Fenestrated System is placed.
  Interventions: Device: Endovascular Aortic Aneurysm Repair (Endologix Fenestrated Stent Graft System)

INTERVENTIONS:
Device: Endovascular Aortic Aneurysm Repair (Endologix Fenestrated Stent Graft System) — Endovascular repair of juxtarenal or pararenal aortic aneurysm using the Endologix Fenestrated Stent Graft System
  Other Names: Ventana; Xpand

SUMMARY:
The aim of this study is to evaluate the safety and feasibility of the Endologix Fenestrated Stent Graft System for the endovascular repair of juxtarenal or pararenal aortic aneurysms.

DETAILED DESCRIPTION:
The Endologix Fenestrated Stent Graft System that will be used in this study has three components, listed below:

1. Endologix unibody bifurcated stent graft
2. Endologix fenestrated proximal extension stent graft
3. Endologix renal stent graft

ELIGIBILITY:
Inclusion Criteria:

* Adequate iliac/femoral access compatible with the required delivery systems
* Non-aneurysmal infrarenal aortic neck <15mm in length
* Most caudal renal artery to aortoiliac bifurcation length >= 70
* SMA to aortoiliac bifurcation length >=90mm
* Proximal non-aneurysmal aortic neck below the SMA with diameter 18 to 34 mm, length >=15mm and angle <=60° to the aneurysm sac
* Angle <=60° (clock face) between the SMA and CA
* Renal arteries both at or below the SMA by <=35mm and within 30mm of each other axially, with 4 to 8mm lumen diameter, and with clockface angle of 90° to 210° to each other
* Common iliac artery distal fixation site with: distal fixation length >=15mm, with diameter >=10 mm and <=23 mm and angle <=90° to the aortic bifurcation
* Ability to preserve at least one hypogastric artery

Exclusion Criteria:

* Life expectancy <2 years as judged by the investigator
* Psychiatric or other condition that may interfere with the study
* Participating in the enrollment or 30-day follow-up phase of another clinical study
* Known allergy to any device component
* Coagulopathy or uncontrolled bleeding disorder
* Contraindication to contrast media or anticoagulants
* Ruptured, leaking, or mycotic aneurysm
* Aortic dissection Serum creatinine (S-Cr) level >2.0 mg/dL
* Traumatic vascular injury
* Active systemic or localized groin infection
* Connective tissue disease (e.g., Marfan's Syndrome)
* Recent(within prior three months)cerebrovascular accident
* Recent(within prior three months)myocardial infarction
* Prior renal transplant
* Length of either renal artery to be stented <12mm
* Significant occlusive disease or calcification of either renal artery (>70%)
* An essential accessory renal artery
* Indispensable inferior mesenteric artery
* Untreated aneurysmal disease of the descending thoracic aorta
* Clinically significant mural thrombus circumferentially in the suprarenal segment
* Prior iliac artery stent implanted that may interfere with delivery system introduction
* Unsuitable vascular anatomy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-10-19 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2018-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clair, MD, Principal Investigator — The Cleveland Clinic; Andrew Holden, MD, Principal Investigator — Auckland City Hospital; Renato Mertens, MD, Principal Investigator — Hospital Universidad Catolica
Locations (8):
- United States (3):
  - UCLA, Los Angeles, California
  - University of Indiana, Indianapolis, Indiana
  - Cleveland Clinic Foundation, Cleveland, Ohio
- Hospital Universidad Catolica, Santiago, Chile
- Bureau de Recherche Clinique, Créteil, France
- Rijnstate Hospital, Arnhem, Netherlands
- Auckland City Hospital, Auckland, New Zealand
- St. George's Vascular Institute, London, United Kingdom

REFERENCES:
- [Derived] Mertens R, Bergoeing M, Marine L, Valdes F, Kramer A, Vergara J. Ventana fenestrated stent-graft system for endovascular repair of juxtarenal aortic aneurysms. J Endovasc Ther. 2012 Apr;19(2):173-8. doi: 10.1583/11-3706.1. PMID 22545881

RESULTS

PARTICIPANT FLOW:
Groups:
- Ventana Fenestrated System: All patients meet study criteria receives a single use Ventana Fenestrated System, which requires administration of intravascular contrast. Catheter advancement is performed under fluoroscopic guidance and Ventana Fenestrated System is placed.
  Endovascular Aortic Aneurysm Repair (Endologix Fenestrated Stent Graft System): Endovascular repair of juxtarenal or pararenal aortic aneurysm using the Endologix Fenestrated Stent Graft System
Period: Overall Study
Arm/Group | Ventana Fenestrated System
Started | 49
Completed | 16
Not Completed | 33
Not completed — Death | 20
Not completed — Withdrawals/Lost to Follow-up | 10
Not completed — Conversion | 2
Not completed — missed visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 14
  Netherlands | 5
  United States | 4
  United Kingdom | 6
  Chile | 11
  France | 9
ASA Class 3 or 4 [Count of Participants; unit: Participants] — ASA (American society of anesthesiologists) classifications explained below:
  ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  Participants | 28
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.1 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint
Description: Major adverse events defined as:
  * All-cause death
  * Bowel ischemia
  * Myocardial infarction
  * Paraplegia
  * Renal failure
  * Respiratory failure
  * Stroke
  * Blood loss >=1,000cc
Time Frame: 30 days
Measure: Number; unit: events
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
events
  All Cause Death | 0
  Bowel Ischemia | 0
  Myocardial Infarction | 0
  Paraplegia | 1
  Procedural Blood Loss | 7
  Renal Failure 1 - Temp/Perm Hemodialysis | 2
  Renal Failure 2 - Serum Creat rise > 0.5mg/dL | 0
  Respiratory Failure 1 - Pneumonia | 0
  Stroke | 0

2. Secondary Outcome: Feasibility/Effectiveness
Description: Successful device delivery and deployment with patency of the renal and aortic endografts without Type I/III endoleak.
  1. Treatment Success is defined as procedural technical success with device patency and the absence of type I/III endoleak
  2. Procedural Technical Success is defined as a subject with successful implant.
  3. Aneurysm Rupture: An aneurysm is a balloon-like bulge of an artery wall. As an aneurysm grows it puts pressure on nearby structures and may eventually rupture.
  4. Clinically Significant Device Migration: Core Lab reported aortic stent graft movement >10mm
  5. Type I/III/IV Endoleak: Core Lab reported endoleak: between the endograft and the vessel either at the proximal attachment point (Type IA), or at the distal attachment point (Type IB), or between endograft components (Type III) or transgraft (Type IV).
  6. Type II Endoleak: Core Lab reported endoleak emanating from a patent collateral vessel (e.g., inferior mesenteric artery, lumbar artery).
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Participants
  Treatment Success | 31
  Unsuccessful Treatment | 18
  Procedural Technical Success | 47
  Aneurysm Rupture | 1
  Conversion to open repair | 1
  Secondary Interventions | 13
  Aneurysm Enlargement | 3
  Clinically Significant Migration | 1
  Type IA Endoleak | 0
  Type IB Endoleak | 0
  Type IIIA Endoleak | 3
  Type IIIB Endoleak | 2

3. Secondary Outcome: Procedural/In-hospital Evaluations
Description: Fluoroscopy time, Renal Artery Cannulation time and procedure time
Time Frame: Procedurally and to hospital discharge
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
minutes
  Fluoroscopy Time | 58 (37)
  Renal Artery Cannulation Time | 51 (57)
  Total Procedure Time | 202 (72)

4. Secondary Outcome: Mortality
Description: All-cause and aneurysm-related
Time Frame: Procedurally and to 5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Participants
  All Cause Deaths | 20
  Aneurysm Related Deaths | 5

5. Secondary Outcome: Major Adverse Events
Description: All-cause mortality, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, stroke, blood loss >1,000cc
Time Frame: >30 Days to 5 Years
Measure: Number; unit: Number of events
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Number of events
  All Cause Death | 6
  Bowel Ischemia | 0
  Myocardial Infarction | 2
  Paraplegia | 0
  Procedural Blood loss | 0
  Renal Failure 1 - Temp/Perm Hemodialysis | 4
  Renal Failure 2 - Serum Creat rise >0.5mg/dL | 1
  Respiratory Failure 1 - Pneumonia | 2
  Stroke | 0

6. Secondary Outcome: Number of Participants With Renal Dysfunction
Description: Renal Dysfunction, Renal Dysfunction In subjects with baseline eGFR>=60 and Renal Dysfunction In subjects with baseline eGFR <60
Time Frame: 30 Days, 6 Months and Years 1 to 5
Population: All available data has been reported
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Participants
  Renal Dysfunction-1 Month: number analyzed (Participants) | 40
  Renal Dysfunction-1 Month | 4
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 1 Month: number analyzed (Participants) | 21
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 1 Month | 2
  Renal Dysfunction in subjects with Baseline eGFR <60 - 1 Month: number analyzed (Participants) | 19
  Renal Dysfunction in subjects with Baseline eGFR <60 - 1 Month | 2
  Renal Dysfunction-6 Month: number analyzed (Participants) | 42
  Renal Dysfunction-6 Month | 9
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 6 Month: number analyzed (Participants) | 24
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 6 Month | 5
  Renal Dysfunction in subjects with Baseline eGFR <60 - 6 Month: number analyzed (Participants) | 18
  Renal Dysfunction in subjects with Baseline eGFR <60 - 6 Month | 4
  Renal Dysfunction-1 Year: number analyzed (Participants) | 40
  Renal Dysfunction-1 Year | 13
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 1 Year: number analyzed (Participants) | 24
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 1 Year | 7
  Renal Dysfunction in subjects with Baseline eGFR <60 - 1 Year: number analyzed (Participants) | 16
  Renal Dysfunction in subjects with Baseline eGFR <60 - 1 Year | 6
  Renal Dysfunction- 2 Year: number analyzed (Participants) | 36
  Renal Dysfunction- 2 Year | 7
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 2 Year: number analyzed (Participants) | 23
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 2 Year | 4
  Renal Dysfunction in subjects with Baseline eGFR <60 - 2 Year: number analyzed (Participants) | 13
  Renal Dysfunction in subjects with Baseline eGFR <60 - 2 Year | 3
  Renal Dysfunction- 3 Year: number analyzed (Participants) | 20
  Renal Dysfunction- 3 Year | 5
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 3 Year: number analyzed (Participants) | 14
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 3 Year | 3
  Renal Dysfunction in subjects with Baseline eGFR <60 - 3 Year: number analyzed (Participants) | 6
  Renal Dysfunction in subjects with Baseline eGFR <60 - 3 Year | 2
  Renal Dysfunction-4 Year: number analyzed (Participants) | 16
  Renal Dysfunction-4 Year | 3
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 4 Year: number analyzed (Participants) | 10
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 4 Year | 2
  Renal Dysfunction in subjects with Baseline eGFR <60 - 4 Year: number analyzed (Participants) | 6
  Renal Dysfunction in subjects with Baseline eGFR <60 - 4 Year | 1
  Renal Dysfunction- 5 Year: number analyzed (Participants) | 14
  Renal Dysfunction- 5 Year | 4
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 5 Year: number analyzed (Participants) | 9
  Renal Dysfunction in subjects with Baseline eGFR >=60 - 5 Year | 2
  Renal Dysfunction in subjects with Baseline eGFR <60 - 5 Year: number analyzed (Participants) | 5
  Renal Dysfunction in subjects with Baseline eGFR <60 - 5 Year | 2

7. Secondary Outcome: Aneurysm Rupture
Description: Internal bleeding or leaking of blood from the aneurysm subsequent to the index procedure
Time Frame: Procedurally and to 5 Years
Population: All available data has been reported
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Participants
  Aneurysm rupture within 30 days | 0
  Aneurysm rupture 30 days- 1 Year | 0
  Aneurysm rupture 1-2 Years: number analyzed (Participants) | 42
  Aneurysm rupture 1-2 Years | 1
  Aneurysm rupture 2-3 Years: number analyzed (Participants) | 39
  Aneurysm rupture 2-3 Years | 2
  Aneurysm rupture 3-4 Years: number analyzed (Participants) | 28
  Aneurysm rupture 3-4 Years | 0
  Aneurysm rupture 4-5 Years: number analyzed (Participants) | 20
  Aneurysm rupture 4-5 Years | 1

8. Secondary Outcome: Conversion to Open Repair
Description: Open surgical repair of the aortic aneurysm due to unsuccessful delivery or deployment of the stent graft, due to complications or other clinical situations that precluded successful endovascular treatment, or at any time following initial successful endovascular treatment for any reason
Time Frame: Procedurally and to 5 Years
Population: All available data has been reported
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Participants
  Open repair within 30 days | 0
  Open repair 30 days - 1 Year | 0
  Open repair 1 -2 Years: number analyzed (Participants) | 42
  Open repair 1 -2 Years | 0
  Open repair 2 -3 Years: number analyzed (Participants) | 39
  Open repair 2 -3 Years | 1
  Open repair 3-4 Years: number analyzed (Participants) | 28
  Open repair 3-4 Years | 1
  Open repair 4-5 Years: number analyzed (Participants) | 20
  Open repair 4-5 Years | 0

9. Secondary Outcome: Device Integrity
Description: Device Migration, Ventana Stent Fracture, Left renal stent fracture, right renal stent fracture, stent Kinking/Compression
Time Frame: 30 Days, 6 Months, and Years 1 to 5
Population: All data has been entered
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Participants
  Ventana Stent Fracture - 1 Month: number analyzed (Participants) | 29
  Ventana Stent Fracture - 1 Month | 0
  Left Renal Stent Fracture - 1 Month: number analyzed (Participants) | 29
  Left Renal Stent Fracture - 1 Month | 1
  Right Renal Stent Fracture - 1 Month: number analyzed (Participants) | 29
  Right Renal Stent Fracture - 1 Month | 0
  Stent Kinking/Compression - 1 Month: number analyzed (Participants) | 46
  Stent Kinking/Compression - 1 Month | 0
  Device Migration - 6 Month: number analyzed (Participants) | 38
  Device Migration - 6 Month | 1
  Ventana Stent Fracture - 6 Month: number analyzed (Participants) | 30
  Ventana Stent Fracture - 6 Month | 1
  Left Renal Stent Fracture - 6 Month: number analyzed (Participants) | 30
  Left Renal Stent Fracture - 6 Month | 2
  Right Renal Stent Fracture - 6 Month: number analyzed (Participants) | 30
  Right Renal Stent Fracture - 6 Month | 3
  Stent Kinking/Compression - 6 Month: number analyzed (Participants) | 41
  Stent Kinking/Compression - 6 Month | 1
  Device Migration - 1 Year: number analyzed (Participants) | 37
  Device Migration - 1 Year | 0
  Ventana Stent Fracture - 1 Year: number analyzed (Participants) | 30
  Ventana Stent Fracture - 1 Year | 3
  Left Renal Stent Fracture - 1 Year: number analyzed (Participants) | 30
  Left Renal Stent Fracture - 1 Year | 2
  Right Renal Stent Fracture - 1 Year: number analyzed (Participants) | 30
  Right Renal Stent Fracture - 1 Year | 3
  Stent Kinking/Compression - 1 Year: number analyzed (Participants) | 37
  Stent Kinking/Compression - 1 Year | 0
  Device Migration - 2 Year: number analyzed (Participants) | 36
  Device Migration - 2 Year | 0
  Ventana Stent Fracture - 2 Year: number analyzed (Participants) | 27
  Ventana Stent Fracture - 2 Year | 3
  Left Renal Stent Fracture - 2 Year: number analyzed (Participants) | 27
  Left Renal Stent Fracture - 2 Year | 2
  Right Renal Stent Fracture - 2 Year: number analyzed (Participants) | 27
  Right Renal Stent Fracture - 2 Year | 5
  Stent Kinking/Compression - 2 Year: number analyzed (Participants) | 36
  Stent Kinking/Compression - 2 Year | 2
  Device Migration - 3 Year: number analyzed (Participants) | 21
  Device Migration - 3 Year | 0
  Ventana Stent Fracture - 3 Year: number analyzed (Participants) | 17
  Ventana Stent Fracture - 3 Year | 4
  Left Renal Stent Fracture - 3 Year: number analyzed (Participants) | 17
  Left Renal Stent Fracture - 3 Year | 1
  Right Renal Stent Fracture - 3 Year: number analyzed (Participants) | 17
  Right Renal Stent Fracture - 3 Year | 2
  Stent Kinking/Compression - 3 Year: number analyzed (Participants) | 22
  Stent Kinking/Compression - 3 Year | 0
  Device Migration - 4 Year: number analyzed (Participants) | 16
  Device Migration - 4 Year | 0
  Ventana Stent Fracture - 4 Year: number analyzed (Participants) | 15
  Ventana Stent Fracture - 4 Year | 4
  Left Renal Stent Fracture - 4 Year: number analyzed (Participants) | 15
  Left Renal Stent Fracture - 4 Year | 2
  Right Renal Stent Fracture - 4 Year: number analyzed (Participants) | 15
  Right Renal Stent Fracture - 4 Year | 2
  Stent Kinking/Compression - 4 Year: number analyzed (Participants) | 16
  Stent Kinking/Compression - 4 Year | 0
  Device Migration - 5 Year: number analyzed (Participants) | 13
  Device Migration - 5 Year | 0
  Ventana Stent Fracture - 5 Year: number analyzed (Participants) | 11
  Ventana Stent Fracture - 5 Year | 4
  Left Renal Stent Fracture - 5 Year: number analyzed (Participants) | 11
  Left Renal Stent Fracture - 5 Year | 1
  Right Renal Stent Fracture - 5 Year: number analyzed (Participants) | 11
  Right Renal Stent Fracture - 5 Year | 2
  Stent Kinking/Compression - 5 Year: number analyzed (Participants) | 13
  Stent Kinking/Compression - 5 Year | 0

10. Secondary Outcome: Stent Graft Patency
Description: Ventana and Bifurcated occlusion, LRA (Left renal artery) occlusion and RRA (right renal artery) occlusion
Time Frame: 30 Days, 6 Months, and Years 1 to 5
Population: All available data has been entered.
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Participants
  Ventana and Bifurcated occlusion - 1 Month: number analyzed (Participants) | 45
  Ventana and Bifurcated occlusion - 1 Month | 0
  LRA Occlusion - 1 Month: number analyzed (Participants) | 45
  LRA Occlusion - 1 Month | 0
  RRA Occlusion - 1 Month: number analyzed (Participants) | 45
  RRA Occlusion - 1 Month | 0
  Ventana and Bifurcated Occlusion - 6 Month: number analyzed (Participants) | 40
  Ventana and Bifurcated Occlusion - 6 Month | 0
  LRA Occlusion - 6 Month: number analyzed (Participants) | 40
  LRA Occlusion - 6 Month | 1
  RRA Occlusion - 6 Month: number analyzed (Participants) | 40
  RRA Occlusion - 6 Month | 1
  Ventana and Bifurcated occlusion - 1 Year: number analyzed (Participants) | 35
  Ventana and Bifurcated occlusion - 1 Year | 1
  LRA Occlusion - 1 Year: number analyzed (Participants) | 35
  LRA Occlusion - 1 Year | 1
  RRA Occlusion - 1 Year: number analyzed (Participants) | 35
  RRA Occlusion - 1 Year | 1
  Ventana and Bifurcated occlusion - 2 Year: number analyzed (Participants) | 35
  Ventana and Bifurcated occlusion - 2 Year | 1
  LRA Occlusion - 2 Year: number analyzed (Participants) | 35
  LRA Occlusion - 2 Year | 4
  RRA Occlusion - 2 Year: number analyzed (Participants) | 35
  RRA Occlusion - 2 Year | 1
  Ventana and Bifurcated occlusion - 3 Year: number analyzed (Participants) | 21
  Ventana and Bifurcated occlusion - 3 Year | 0
  LRA Occlusion - 3 Year: number analyzed (Participants) | 21
  LRA Occlusion - 3 Year | 1
  RRA Occlusion - 3 Year: number analyzed (Participants) | 21
  RRA Occlusion - 3 Year | 0
  Ventana and Bifurcated occlusion - 4 Year: number analyzed (Participants) | 16
  Ventana and Bifurcated occlusion - 4 Year | 0
  LRA Occlusion - 4 Year: number analyzed (Participants) | 16
  LRA Occlusion - 4 Year | 1
  RRA Occlusion - 4 Year: number analyzed (Participants) | 16
  RRA Occlusion - 4 Year | 0
  Ventana and Bifurcated occlusion - 5 Year: number analyzed (Participants) | 13
  Ventana and Bifurcated occlusion - 5 Year | 0
  LRA Occlusion - 5 Year: number analyzed (Participants) | 13
  LRA Occlusion - 5 Year | 2
  RRA Occlusion - 5 Year: number analyzed (Participants) | 13
  RRA Occlusion - 5 Year | 1

11. Secondary Outcome: Aneurysm Diameter Change
Description: Change in aneurysm sac diameter - decrease > 5mm, Increase > 5mm, Stable (+/- 5mm) and No growth.
Time Frame: 6 Months, and Years 1 to 5
Population: All data has been entered
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Participants
  Decrease (>5mm)- 6 Month: number analyzed (Participants) | 39
  Decrease (>5mm)- 6 Month | 4
  Increase (>5mm) - 6 Month: number analyzed (Participants) | 39
  Increase (>5mm) - 6 Month | 1
  Stable (±5mm) - 6 Month: number analyzed (Participants) | 39
  Stable (±5mm) - 6 Month | 34
  No Growth - 6 Month: number analyzed (Participants) | 39
  No Growth - 6 Month | 38
  Decrease (>5mm)- 1 Year: number analyzed (Participants) | 35
  Decrease (>5mm)- 1 Year | 7
  Increase (>5mm) - 1 Year: number analyzed (Participants) | 35
  Increase (>5mm) - 1 Year | 0
  Stable (±5mm) - 1 Year: number analyzed (Participants) | 35
  Stable (±5mm) - 1 Year | 28
  No Growth - 1 Year: number analyzed (Participants) | 35
  No Growth - 1 Year | 35
  Decrease (>5mm)- 2 Year: number analyzed (Participants) | 35
  Decrease (>5mm)- 2 Year | 9
  Increase (>5mm) - 2 Year: number analyzed (Participants) | 35
  Increase (>5mm) - 2 Year | 8
  Stable (±5mm) - 2 Year: number analyzed (Participants) | 35
  Stable (±5mm) - 2 Year | 18
  No Growth - 2 Year: number analyzed (Participants) | 35
  No Growth - 2 Year | 27
  Decrease (>5mm)- 3 Year: number analyzed (Participants) | 22
  Decrease (>5mm)- 3 Year | 8
  Increase (>5mm) - 3 Year: number analyzed (Participants) | 22
  Increase (>5mm) - 3 Year | 1
  Stable (±5mm) - 3 Year: number analyzed (Participants) | 22
  Stable (±5mm) - 3 Year | 13
  No Growth - 3 Year: number analyzed (Participants) | 22
  No Growth - 3 Year | 21
  Decrease (>5mm)- 4 Year: number analyzed (Participants) | 16
  Decrease (>5mm)- 4 Year | 6
  Increase (>5mm) - 4 Year: number analyzed (Participants) | 16
  Increase (>5mm) - 4 Year | 0
  Stable (±5mm) - 4 Year: number analyzed (Participants) | 16
  Stable (±5mm) - 4 Year | 10
  No Growth - 4 Year: number analyzed (Participants) | 16
  No Growth - 4 Year | 16
  Decrease (>5mm)- 5 Year: number analyzed (Participants) | 13
  Decrease (>5mm)- 5 Year | 4
  Increase (>5mm) - 5 Year: number analyzed (Participants) | 13
  Increase (>5mm) - 5 Year | 4
  Stable (±5mm) - 5 Year: number analyzed (Participants) | 13
  Stable (±5mm) - 5 Year | 5
  No Growth - 5 Year: number analyzed (Participants) | 13
  No Growth - 5 Year | 9

12. Secondary Outcome: Secondary Procedures
Description: Non-diagnostic intervention after the index procedure intended to correct or repair an endoleak (device-related: Type I (proximal or distal), Type III, Type IV; non-device related: Type II), device migration, or other device defect.
Time Frame: 30 Days, 6 Month and Years 1 to 5
Population: All data has been entered
Measure: Count of Participants; unit: Participants
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
Participants
  Aneurysm Expansion - Conversion to open repair - 30 days | 0
  Aneurysm Expansion - Conversion to open repair - 6 Month | 0
  Aneurysm Expansion - Conversion to open repair - 1 Year | 0
  Aneurysm Expansion - Conversion to open repair - 2 Year: number analyzed (Participants) | 42
  Aneurysm Expansion - Conversion to open repair - 2 Year | 0
  Aneurysm Expansion - Conversion to open repair - 3 Year: number analyzed (Participants) | 39
  Aneurysm Expansion - Conversion to open repair - 3 Year | 0
  Aneurysm Expansion - Conversion to open repair - 4 Year: number analyzed (Participants) | 28
  Aneurysm Expansion - Conversion to open repair - 4 Year | 1
  Aneurysm Expansion - Conversion to open repair - 5 Year: number analyzed (Participants) | 20
  Aneurysm Expansion - Conversion to open repair - 5 Year | 0
  Aneurysm Rupture - Conversion to open repair - 30 days | 0
  Aneurysm Rupture - Conversion to open repair - 6 Month | 0
  Aneurysm Rupture - Conversion to open repair - 1 Year | 0
  Aneurysm Rupture - Conversion to open repair - 2 Year: number analyzed (Participants) | 42
  Aneurysm Rupture - Conversion to open repair - 2 Year | 1
  Aneurysm Rupture - Conversion to open repair - 3 Year: number analyzed (Participants) | 39
  Aneurysm Rupture - Conversion to open repair - 3 Year | 0
  Aneurysm Rupture - Conversion to open repair - 4 Year: number analyzed (Participants) | 28
  Aneurysm Rupture - Conversion to open repair - 4 Year | 0
  Aneurysm Rupture - Conversion to open repair - 5 Year: number analyzed (Participants) | 20
  Aneurysm Rupture - Conversion to open repair - 5 Year | 0
  Aortic Occlusion -Bypass - Other- 30 Days | 0
  Aortic Occlusion -Bypass - Other- 6 Month | 0
  Aortic Occlusion -Bypass - Other- 1 Year | 0
  Aortic Occlusion -Bypass - Other- 2 Year: number analyzed (Participants) | 42
  Aortic Occlusion -Bypass - Other- 2 Year | 1
  Aortic Occlusion -Bypass - Other- 3 Year: number analyzed (Participants) | 39
  Aortic Occlusion -Bypass - Other- 3 Year | 0
  Aortic Occlusion -Bypass - Other- 4 Year: number analyzed (Participants) | 28
  Aortic Occlusion -Bypass - Other- 4 Year | 0
  Aortic Occlusion -Bypass - Other- 5 Year: number analyzed (Participants) | 20
  Aortic Occlusion -Bypass - Other- 5 Year | 0
  Device Migration - Renal Stenting - 30 Days | 0
  Device Migration - Renal Stenting - 6 Month | 0
  Device Migration - Renal Stenting - 1 Year | 0
  Device Migration - Renal Stenting - 2 Year: number analyzed (Participants) | 42
  Device Migration - Renal Stenting - 2 Year | 1
  Device Migration - Renal Stenting - 3 Year: number analyzed (Participants) | 39
  Device Migration - Renal Stenting - 3 Year | 0
  Device Migration - Renal Stenting 4 Year: number analyzed (Participants) | 28
  Device Migration - Renal Stenting 4 Year | 0
  Device Migration - Renal Stenting - 5 Year: number analyzed (Participants) | 20
  Device Migration - Renal Stenting - 5 Year | 0
  Iliac Artery Stenosis/Occlusion - 30 Days | 2
  Iliac Artery Stenosis/Occlusion - 6 Month | 1
  Iliac Artery Stenosis/Occlusion - 1 Year | 3
  Iliac Artery Stenosis/Occlusion - 2 Year: number analyzed (Participants) | 42
  Iliac Artery Stenosis/Occlusion - 2 Year | 0
  Iliac Artery Stenosis/Occlusion - 3 Year: number analyzed (Participants) | 39
  Iliac Artery Stenosis/Occlusion - 3 Year | 0
  Iliac Artery Stenosis/Occlusion - 4 Year: number analyzed (Participants) | 28
  Iliac Artery Stenosis/Occlusion - 4 Year | 0
  Iliac Artery Stenosis/Occlusion - 5 Year: number analyzed (Participants) | 20
  Iliac Artery Stenosis/Occlusion - 5 Year | 0
  Renal Artery Stenosis/Occlusion - 30 Days | 0
  Renal Artery Stenosis/Occlusion - 6 Month | 9
  Renal Artery Stenosis/Occlusion - 1 Year | 9
  Renal Artery Stenosis/Occlusion - 2 Year: number analyzed (Participants) | 42
  Renal Artery Stenosis/Occlusion - 2 Year | 2
  Renal Artery Stenosis/Occlusion - 3 Year: number analyzed (Participants) | 39
  Renal Artery Stenosis/Occlusion - 3 Year | 0
  Renal Artery Stenosis/Occlusion - 4 Year: number analyzed (Participants) | 28
  Renal Artery Stenosis/Occlusion - 4 Year | 0
  Renal Artery Stenosis/Occlusion - 5 Year: number analyzed (Participants) | 20
  Renal Artery Stenosis/Occlusion - 5 Year | 0
  SMA Artery Occlusion- 30 Days | 1
  SMA Artery Occlusion- 6 Month | 0
  SMA Artery Occlusion- 1 Year | 1
  SMA Artery Occlusion- 2 Year: number analyzed (Participants) | 42
  SMA Artery Occlusion- 2 Year | 0
  SMA Artery Occlusion- 3 Year: number analyzed (Participants) | 39
  SMA Artery Occlusion- 3 Year | 0
  SMA Artery Occlusion- 4 Year: number analyzed (Participants) | 28
  SMA Artery Occlusion- 4 Year | 0
  SMA Artery Occlusion- 5 Year: number analyzed (Participants) | 20
  SMA Artery Occlusion- 5 Year | 0
  Stent Fracture - 30 Days | 0
  Stent Fracture - 6 Month | 0
  Stent Fracture - 1 Year | 0
  Stent Fracture - 2 Year: number analyzed (Participants) | 42
  Stent Fracture - 2 Year | 1
  Stent Fracture - 3 Year: number analyzed (Participants) | 39
  Stent Fracture - 3 Year | 2
  Stent Fracture - 4 Year: number analyzed (Participants) | 28
  Stent Fracture - 4 Year | 1
  Stent Fracture - 5 Year: number analyzed (Participants) | 20
  Stent Fracture - 5 Year | 0
  Stent Migration - 30 Days | 0
  Stent Migration - 6 Month | 0
  Stent Migration - 1 Year | 0
  Stent Migration - 2 Year: number analyzed (Participants) | 42
  Stent Migration - 2 Year | 0
  Stent Migration - 3 Year: number analyzed (Participants) | 39
  Stent Migration - 3 Year | 0
  Stent Migration - 4 Year: number analyzed (Participants) | 28
  Stent Migration - 4 Year | 0
  Stent Migration - 5 Year: number analyzed (Participants) | 20
  Stent Migration - 5 Year | 1
  Type IA Endoleak - 30 Days | 0
  Type IA Endoleak - 6 Month | 1
  Type IA Endoleak - 1 Year | 1
  Type IA Endoleak - 2 Year: number analyzed (Participants) | 42
  Type IA Endoleak - 2 Year | 0
  Type IA Endoleak - 3 Year: number analyzed (Participants) | 39
  Type IA Endoleak - 3 Year | 0
  Type IA Endoleak - 4 Year: number analyzed (Participants) | 28
  Type IA Endoleak - 4 Year | 0
  Type IA Endoleak - 5 Year: number analyzed (Participants) | 20
  Type IA Endoleak - 5 Year | 0
  Liquid Embolization - 30 Days | 0
  Liquid Embolization - 6 Month | 1
  Liquid Embolization - 1 Year | 1
  Liquid Embolization - 2 Year: number analyzed (Participants) | 42
  Liquid Embolization - 2 Year | 0
  Liquid Embolization - 3 Year: number analyzed (Participants) | 39
  Liquid Embolization - 3 Year | 0
  Liquid Embolization - 4 Year: number analyzed (Participants) | 28
  Liquid Embolization - 4 Year | 0
  Liquid Embolization - 5 Year: number analyzed (Participants) | 20
  Liquid Embolization - 5 Year | 0
  Type IB Endoleak - 30 Days | 0
  Type IB Endoleak - 6 Month | 0
  Type IB Endoleak - 1 Year | 0
  Type IB Endoleak - 2 Year: number analyzed (Participants) | 42
  Type IB Endoleak - 2 Year | 0
  Type IB Endoleak - 3 Year: number analyzed (Participants) | 39
  Type IB Endoleak - 3 Year | 1
  Type IB Endoleak - 4 Year: number analyzed (Participants) | 28
  Type IB Endoleak - 4 Year | 0
  Type IB Endoleak - 5 Year: number analyzed (Participants) | 20
  Type IB Endoleak - 5 Year | 0
  Conversion to Open Repair - 30 Days | 0
  Conversion to Open Repair - 6 Month | 0
  Conversion to Open Repair - 1 Year | 0
  Conversion to Open Repair - 2 Year: number analyzed (Participants) | 42
  Conversion to Open Repair - 2 Year | 0
  Conversion to Open Repair - 3 Year: number analyzed (Participants) | 39
  Conversion to Open Repair - 3 Year | 1
  Conversion to Open Repair - 4 Year: number analyzed (Participants) | 28
  Conversion to Open Repair - 4 Year | 0
  Conversion to Open Repair - 5 Year: number analyzed (Participants) | 20
  Conversion to Open Repair - 5 Year | 0
  Type II Endoleak - 30 Days | 0
  Type II Endoleak - 6 Month | 0
  Type II Endoleak - 1 Year | 0
  Type II Endoleak - 2 Year: number analyzed (Participants) | 42
  Type II Endoleak - 2 Year | 1
  Type II Endoleak - 3 Year: number analyzed (Participants) | 39
  Type II Endoleak - 3 Year | 1
  Type II Endoleak - 4 Year: number analyzed (Participants) | 28
  Type II Endoleak - 4 Year | 0
  Type II Endoleak - 5 Year: number analyzed (Participants) | 20
  Type II Endoleak - 5 Year | 0
  Coil Embolization - 30 Days | 0
  Coil Embolization - 6 Month | 0
  Coil Embolization - 1 Year | 0
  Coil Embolization - 2 Year: number analyzed (Participants) | 42
  Coil Embolization - 2 Year | 1
  Coil Embolization - 3 Year: number analyzed (Participants) | 39
  Coil Embolization - 3 Year | 1
  Coil Embolization - 4 Year: number analyzed (Participants) | 28
  Coil Embolization - 4 Year | 0
  Coil Embolization - 5 Year: number analyzed (Participants) | 20
  Coil Embolization - 5 Year | 0
  Type III Endoleak - 30 Days | 1
  Type III Endoleak - 6 Month | 1
  Type III Endoleak - 1 Year | 2
  Type III Endoleak - 2 Year: number analyzed (Participants) | 42
  Type III Endoleak - 2 Year | 2
  Type III Endoleak - 3 Year: number analyzed (Participants) | 39
  Type III Endoleak - 3 Year | 4
  Type III Endoleak - 4 Year: number analyzed (Participants) | 28
  Type III Endoleak - 4 Year | 0
  Type III Endoleak - 5 Year: number analyzed (Participants) | 20
  Type III Endoleak - 5 Year | 1
  Aortic Extension- 30 Days | 0
  Aortic Extension- 6 Month | 0
  Aortic Extension- 1 Year | 0
  Aortic Extension- 2 Year: number analyzed (Participants) | 42
  Aortic Extension- 2 Year | 1
  Aortic Extension- 3 Year: number analyzed (Participants) | 39
  Aortic Extension- 3 Year | 2
  Aortic Extension- 4 Year: number analyzed (Participants) | 28
  Aortic Extension- 4 Year | 0
  Aortic Extension- 5 Year: number analyzed (Participants) | 20
  Aortic Extension- 5 Year | 0
  Aortic Revision - 30 Days | 0
  Aortic Revision - 6 Month | 1
  Aortic Revision - 1 Year | 1
  Aortic Revision - 2 Year: number analyzed (Participants) | 42
  Aortic Revision - 2 Year | 1
  Aortic Revision - 3 Year: number analyzed (Participants) | 39
  Aortic Revision - 3 Year | 2
  Aortic Revision - 4 Year: number analyzed (Participants) | 28
  Aortic Revision - 4 Year | 0
  Aortic Revision - 5 Year: number analyzed (Participants) | 20
  Aortic Revision - 5 Year | 1
  Balloon Angioplasty - 30 Days | 1
  Balloon Angioplasty - 6 Month | 0
  Balloon Angioplasty - 1 Year | 1
  Balloon Angioplasty - 2 Year: number analyzed (Participants) | 42
  Balloon Angioplasty - 2 Year | 0
  Balloon Angioplasty - 3 Year: number analyzed (Participants) | 39
  Balloon Angioplasty - 3 Year | 0
  Balloon Angioplasty - 4 Year: number analyzed (Participants) | 28
  Balloon Angioplasty - 4 Year | 0
  Balloon Angioplasty - 5 Year: number analyzed (Participants) | 20
  Balloon Angioplasty - 5 Year | 0
  Iliac Extension - 30 Days | 0
  Iliac Extension - 6 Month | 0
  Iliac Extension - 1 Year | 0
  Iliac Extension - 2 Year: number analyzed (Participants) | 42
  Iliac Extension - 2 Year | 0
  Iliac Extension - 3 Year: number analyzed (Participants) | 39
  Iliac Extension - 3 Year | 0
  Iliac Extension - 4 Year: number analyzed (Participants) | 28
  Iliac Extension - 4 Year | 0
  Iliac Extension - 5 Year: number analyzed (Participants) | 20
  Iliac Extension - 5 Year | 1
  Renal Stenting - 30 Days | 0
  Renal Stenting - 6 Month | 0
  Renal Stenting - 1 Year | 0
  Renal Stenting - 2 Year: number analyzed (Participants) | 42
  Renal Stenting - 2 Year | 1
  Renal Stenting - 3 Year: number analyzed (Participants) | 39
  Renal Stenting - 3 Year | 1
  Renal Stenting - 4 Year: number analyzed (Participants) | 28
  Renal Stenting - 4 Year | 0
  Renal Stenting - 5 Year: number analyzed (Participants) | 20
  Renal Stenting - 5 Year | 0

13. Secondary Outcome: Procedural/In-hospital Evaluations
Description: Contrast volume and estimated blood loss
Time Frame: Procedurally and to hospital discharge
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
mL
  Contrast Volume | 205 (107)
  Blood Loss | 581 (396)

14. Secondary Outcome: Procedural/In-hospital Evaluations
Description: Time to hospital discharge
Time Frame: Discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ventana Fenestrated System
Number analyzed (Participants) | 49
days | 5 (4)

ADVERSE EVENTS:
Time Frame: 5 Years
Arm/Group | Ventana Fenestrated System
All-Cause Mortality (participants affected / at risk) | 20/49
Serious Adverse Events (participants affected / at risk) | 42/49
Other Adverse Events (participants affected / at risk) | 46/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ventana Fenestrated System (N=49)
Arrhythmia (Cardiac disorders) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac ischemia (Cardiac disorders) | 1 (1)
Congestive cardiac failure aggravated (Cardiac disorders) | 3 (4)
Congestive heart failure (Cardiac disorders) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Decompensation cardiac (Cardiac disorders) | 1 (1)
Diastolic heart failure (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Unstable angina (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Bowel ischemia (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal hemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Arterial stent occlusion (General disorders) | 1 (1)
Catheter site hematoma (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Complication of device insertion (General disorders) | 1 (1)
Device dislocation (General disorders) | 1 (2)
Device fracture (General disorders) | 1 (1)
Device misdeployment (General disorders) | 1 (1)
Endoleak (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Multi organ failure (General disorders) | 1 (1)
Multiple organ failure (General disorders) | 1 (1)
Stent dislodgement (General disorders) | 1 (1)
Stent occlusion (General disorders) | 5 (5)
Stent strut fracture (General disorders) | 2 (2)
Stent-graft compression (General disorders) | 1 (1)
Stent-graft endoleak type IA (General disorders) | 1 (1)
Stent-graft endoleak type IB (General disorders) | 1 (2)
Stent-graft endoleak type II (General disorders) | 4 (4)
Stent-graft endoleak type III (General disorders) | 8 (8)
Stent-graft malfunction (General disorders) | 1 (1)
Stent-graft separation (General disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Acute on chronic bronchitis (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Diarrhea, Clostridium difficile (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Graft infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Post procedural site wound infection (Infections and infestations) | 1 (1)
Staphylococcus aureus bacteraemia (Infections and infestations) | 1 (1)
Staphylococcus epidermidis septicemia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 2 (2)
Intraoperative bleeding (Injury, poisoning and procedural complications) | 2 (2)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Angiogram (Investigations) | 1 (1)
Increased serum creatinine (Investigations) | 3 (3)
Vascular imaging (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Loin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenocarcinoma lung stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bowel cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Brain tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer of lung stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Esophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Ischemic stroke (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 2 (2)
Anuria (Renal and urinary disorders) | 1 (1)
Bilateral renal artery stenosis (Renal and urinary disorders) | 1 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Chronic renal failure worsened (Renal and urinary disorders) | 2 (2)
End stage renal failure (Renal and urinary disorders) | 2 (2)
Function kidney decreased (Renal and urinary disorders) | 1 (1)
Kidney dysfunction (Renal and urinary disorders) | 1 (1)
Renal artery occlusion (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Acute on chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 2 (4)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Exacerbation of asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hip arthroplasty (Surgical and medical procedures) | 1 (1)
Intravenous fluids replacement (Surgical and medical procedures) | 1 (3)
Stent removal (Surgical and medical procedures) | 1 (1)
Surgical intervention (Surgical and medical procedures) | 1 (2)
Abdominal aneurysm, ruptured (Vascular disorders) | 3 (3)
Abdominal aortic aneurysm enlargement (Vascular disorders) | 1 (1)
Aneurysm enlargement (Vascular disorders) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 1 (1)
Aortic occlusion (Vascular disorders) | 1 (1)
Arterial bleeding (Vascular disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Arteriovenous graft site stenosis (Vascular disorders) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1)
Femoral artery thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Iliac artery rupture (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ventana Fenestrated System (N=49)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Anemia aggravated (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Acute decompensated heart failure (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Congestive cardiac failure aggravated (Cardiac disorders) | 2 (2)
Congestive heart failure (Cardiac disorders) | 2 (2)
Coronary artery disease aggravated (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 3 (3)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 2 (4)
Visual acuity decreased (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Bowel ischemia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Distended abdomen (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1)
Retroperitoneal hematoma (Gastrointestinal disorders) | 2 (2)
Stomach ulcer with hemorrhage (Gastrointestinal disorders) | 1 (1)
Ankle edema (General disorders) | 1 (1)
Arterial stent occlusion (General disorders) | 2 (2)
Cardiac pacemaker malfunction (General disorders) | 1 (1)
Catheter site hematoma (General disorders) | 4 (4)
Catheter site swelling (General disorders) | 1 (1)
Complication of device insertion (General disorders) | 1 (1)
Debility (General disorders) | 1 (1)
General malaise (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Implant site seroma (General disorders) | 1 (1)
Shivering (General disorders) | 1 (1)
Stent occlusion (General disorders) | 1 (1)
Stent strut fracture (General disorders) | 1 (1)
Stent-graft angulation (General disorders) | 1 (2)
Stent-graft endoleak type II (General disorders) | 6 (6)
Stent-graft endoleak type III (General disorders) | 2 (2)
Stent-graft malfunction (General disorders) | 1 (1)
Stent-graft material failure (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Groin infection (Infections and infestations) | 1 (1)
Infected epidermal cyst (Infections and infestations) | 1 (1)
Infected hydrocele (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary infection (Infections and infestations) | 1 (1)
Anemia postoperative (Injury, poisoning and procedural complications) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Contusion of shoulder region (Injury, poisoning and procedural complications) | 1 (1)
Delirium on emergence (Injury, poisoning and procedural complications) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (2)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative bleeding (Injury, poisoning and procedural complications) | 4 (4)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous hematoma (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Cardiac monitoring (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Creatinine serum increased (Investigations) | 2 (2)
INR increased (Investigations) | 1 (1)
Increased blood pressure (Investigations) | 1 (1)
Increased serum creatinine (Investigations) | 4 (4)
Serum creatinine increased (Investigations) | 1 (1)
Diabetes mellitus loss of control (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Worsening of diabetes (Metabolism and nutrition disorders) | 1 (1)
Acute back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ankle swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hip arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower extremities weakness of (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in thigh (Musculoskeletal and connective tissue disorders) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Larynx carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Abnormal sensation of limbs (Nervous system disorders) | 1 (1)
Carotid occlusion (Nervous system disorders) | 1 (1)
Dementia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
Numbness in leg (Nervous system disorders) | 1 (1)
Palsy Bells (Nervous system disorders) | 1 (1)
Upper limb paresis (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Acute on chronic renal failure (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Chronic renal failure worsened (Renal and urinary disorders) | 1 (3)
Function kidney decreased (Renal and urinary disorders) | 1 (1)
Renal artery dissection (Renal and urinary disorders) | 2 (2)
Renal artery occlusion (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 3 (3)
Renal infarct (Renal and urinary disorders) | 1 (1)
Renal infarction (Renal and urinary disorders) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Blood transfusion (Surgical and medical procedures) | 1 (1)
Abdominal aortic aneurysm enlargement (Vascular disorders) | 2 (2)
Aneurysm enlargement (Vascular disorders) | 1 (1)
Blue toe syndrome (Vascular disorders) | 1 (1)
Claudication (Vascular disorders) | 2 (2)
Groin hematoma (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypertension worsened (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Popliteal artery aneurysm (Vascular disorders) | 1 (1)
Superficial femoral arterial stenosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-03-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT01348828/Prot_SAP_000.pdf
  • Informed Consent Form (2012-01-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT01348828/ICF_001.pdf